CLINICAL TRIAL: NCT02682810
Title: Z 1303 - Point-of-Care Virologic Testing to Improve Outcomes of HIV-Infected Children
Brief Title: Point of Care Virologic Testing to Improve Outcomes of HIV-Infected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 12-1346; 5U01AI100053-03 (NIH)
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-01

CONDITIONS: Early Infant HIV Diagnosis
Keywords: HIV; point-of-care HIV diagnosis; Alere Q; diagnostic; children
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DNA PCR HIV diagnostic test (Active Comparator): SOC or control arm through existing PMTCT program, with DBS samples sent to an off-site laboratory for DNA PCR testing.
  Interventions: Device: DNA PCR HIV diagnostic test
- Alere Q POC nucleic acid-based platform (Experimental): POC test to provide same-day diagnosis
  Interventions: Device: Alere Q

INTERVENTIONS:
Device: DNA PCR HIV diagnostic test — standard of care
  Arms: DNA PCR HIV diagnostic test
Device: Alere Q — POC diagnostic Alere Q qualitative test (along with a DBS drawn for confirmatory DNA PCR)
  Arms: Alere Q POC nucleic acid-based platform

SUMMARY:
This is a two-arm, unmasked, randomized, controlled trial to test the effectiveness of the Alere Q point-of-care (POC) HIV diagnostic assay for use in resource-poor settings.

DETAILED DESCRIPTION:
At public sector clinics in Lusaka, Zambia, approximately 4,000 HIV-exposed infants between 4 and 12 weeks of life will be randomized in this trial of point-of-care virologic testing to improve outcomes of HIV-infected children in Zambia. There is a standard of care (SOC) or control arm and an intervention arm known as the Alere arm. In both study arms, early infant diagnosis (EID) will be provided at 6 weeks of life. Infants randomized to the SOC arm will receive EID through the existing prevention of mother-to-child-transmission (PMTCT) program, with samples sent to an off-site laboratory for DNA PCR testing. Infants randomized to the intervention arm will receive POC diagnostic Alere Q qualitative test (along with a dried blood spot (DBS) drawn for confirmatory DNA PCR).

HIV-infected infants will be followed for 12 months. The acceptability of point-of-care testing for EID will also be determined through the use of cross-sectional surveys of clinicians, laboratory personnel, and parents/guardians.

The feasibility will be assessed by a time-in-motion (TIM) and value stream mapping (VSM) analyses will also be conducted to compare the Alere Q to two additional testing technologies.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 12 weeks of life
* documented HIV exposure through seropositive maternal or infant HIV antibody test
* with a parent or guardian will and able to provide written informed consent and to have the participant followed for 12 months after study enrolment

Exclusion Criteria:

* Infants will be excluded from participation if they have major congenital anomalies or other medical conditions that would require management at a referral facility or otherwise interfere with study procedures

Ages: 4 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4000 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Proportion of HIV-infected children in each arm who remain alive, in care, and with no HIV circulating in their bloodstream 12 months after initial diagnosis | time of initial diagnosis through 12 months post diagnosis

SECONDARY OUTCOMES:
Proportion of HIV-infected children who start anti-retroviral therapy (ART) within 6 months of the initial diagnosis | time of initial diagnosis through 6 months post diagnosis
  Short-term benefit
Proportion of children starting ART who remain in care for 12 months following the initial diagnosis | time of initial diagnostic blood draw through 12 months post diagnosis
  Long-term retention benefit

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Stringer, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (6):
- Zambia (6):
  - Chawama Health Centre, Lusaka
  - Chelstone Health Centre, Lusaka
  - Chilenje Health Centre, Lusaka
  - Chipata Health Centre, Lusaka
  - Kanyama Health Centre, Lusaka
  - Mtendere Health Centre, Lusaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Violari A, Cotton MF, Gibb DM, Babiker AG, Steyn J, Madhi SA, Jean-Philippe P, McIntyre JA; CHER Study Team. Early antiretroviral therapy and mortality among HIV-infected infants. N Engl J Med. 2008 Nov 20;359(21):2233-44. doi: 10.1056/NEJMoa0800971. PMID 19020325
- [Background] UNAIDS. 2014 Progress Report on The Global Plan: http://www.unaids.org/sites/default/files/documents/JC2681_2014-Global-Plan-progress_en.pdf. Accessed: 01 February 2015.
- [Background] Stringer EM, Ekouevi DK, Coetzee D, Tih PM, Creek TL, Stinson K, Giganti MJ, Welty TK, Chintu N, Chi BH, Wilfert CM, Shaffer N, Dabis F, Stringer JS; PEARL Study Team. Coverage of nevirapine-based services to prevent mother-to-child HIV transmission in 4 African countries. JAMA. 2010 Jul 21;304(3):293-302. doi: 10.1001/jama.2010.990. PMID 20639563
- [Background] Stringer JS, Sinkala M, Maclean CC, Levy J, Kankasa C, Degroot A, Stringer EM, Acosta EP, Goldenberg RL, Vermund SH. Effectiveness of a city-wide program to prevent mother-to-child HIV transmission in Lusaka, Zambia. AIDS. 2005 Aug 12;19(12):1309-15. doi: 10.1097/01.aids.0000180102.88511.7d. PMID 16052086
- [Background] Antiretroviral Therapy for HIV Infection in Infants and Children: Towards Universal Access: Recommendations for a Public Health Approach: 2010 Revision. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138576/ PMID 23741772
- [Background] Braun M, Kabue MM, McCollum ED, Ahmed S, Kim M, Aertker L, Chirwa M, Eliya M, Mofolo I, Hoffman I, Kazembe PN, van der Horst C, Kline MW, Hosseinipour MC. Inadequate coordination of maternal and infant HIV services detrimentally affects early infant diagnosis outcomes in Lilongwe, Malawi. J Acquir Immune Defic Syndr. 2011 Apr 15;56(5):e122-8. doi: 10.1097/QAI.0b013e31820a7f2f. PMID 21224736
- [Background] Newell ML, Coovadia H, Cortina-Borja M, Rollins N, Gaillard P, Dabis F; Ghent International AIDS Society (IAS) Working Group on HIV Infection in Women and Children. Mortality of infected and uninfected infants born to HIV-infected mothers in Africa: a pooled analysis. Lancet. 2004 Oct 2-8;364(9441):1236-43. doi: 10.1016/S0140-6736(04)17140-7. PMID 15464184
- [Background] Laursen L. Point-of-care tests poised to alter course of HIV treatment. Nat Med. 2012 Aug;18(8):1156. doi: 10.1038/nm0812-1156. No abstract available. PMID 22869167
- [Background] UNITAID. HIV/AIDS diagnostic technology landscape.Tech. Rep., WHO, Geneva, Switzerland, 2012.
- [Background] Jani IV, Meggi B, Mabunda N, Vubil A, Sitoe NE, Tobaiwa O, Quevedo JI, Lehe JD, Loquiha O, Vojnov L, Peter TF. Accurate early infant HIV diagnosis in primary health clinics using a point-of-care nucleic acid test. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):e1-4. doi: 10.1097/QAI.0000000000000250. PMID 24933096
- [Background] Yusuf S, Collins R, Peto R. Why do we need some large, simple randomized trials? Stat Med. 1984 Oct-Dec;3(4):409-22. doi: 10.1002/sim.4780030421. No abstract available. PMID 6528136
- [Background] Palumbo P, Lindsey JC, Hughes MD, Cotton MF, Bobat R, Meyers T, Bwakura-Dangarembizi M, Chi BH, Musoke P, Kamthunzi P, Schimana W, Purdue L, Eshleman SH, Abrams EJ, Millar L, Petzold E, Mofenson LM, Jean-Philippe P, Violari A. Antiretroviral treatment for children with peripartum nevirapine exposure. N Engl J Med. 2010 Oct 14;363(16):1510-20. doi: 10.1056/NEJMoa1000931. PMID 20942667
- [Background] Bolton-Moore C, Mubiana-Mbewe M, Cantrell RA, Chintu N, Stringer EM, Chi BH, Sinkala M, Kankasa C, Wilson CM, Wilfert CM, Mwango A, Levy J, Abrams EJ, Bulterys M, Stringer JS. Clinical outcomes and CD4 cell response in children receiving antiretroviral therapy at primary health care facilities in Zambia. JAMA. 2007 Oct 24;298(16):1888-99. doi: 10.1001/jama.298.16.1888. PMID 17954540
- [Derived] Chibwesha CJ, Mollan KR, Ford CE, Shibemba A, Saha PT, Lusaka M, Mbewe F, Allmon AG, Lungu R, Spiegel HML, Mweni E, Mwape H, Kankasa C, Chi BH, Stringer JSA. A Randomized Trial of Point-of-Care Early Infant Human Immunodeficiency Virus (HIV) Diagnosis in Zambia. Clin Infect Dis. 2022 Aug 25;75(2):260-268. doi: 10.1093/cid/ciab923. PMID 34718462
- [Derived] Chibwesha CJ, Ford CE, Mollan KR, Stringer JS. Point-of-Care Virologic Testing to Improve Outcomes of HIV-Infected Children in Zambia: A Clinical Trial Protocol. J Acquir Immune Defic Syndr. 2016 Aug 1;72 Suppl 2(Suppl 2):S197-201. doi: 10.1097/QAI.0000000000001050. PMID 27355509
- See also: University of North Carolina website — http://www.unc.edu